CLINICAL TRIAL: NCT04500600
Title: Well-Being and Quality of Life in Cancer Patients and Survivors During the COVID-19 Pandemic
Brief Title: Well-Being and Health-Related Quality of Life in Cancer Patients and Survivors During the COVID-19 Pandemic
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0473; NCI-2020-04604 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0473 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-24; First posted 2020-08-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: COVID-19 Infection; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire): Patients complete an online questionnaire over 10 minutes regarding the COVID-19 pandemic including testing, risks of exposure, whether people they know have acquired COVID-19, as well as questions on how the pandemic has impacted their quality of life.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This study investigates the well-being and health-related quality of life in cancer patients and survivors during the COVID-19 pandemic. Using questionnaires may help researchers gain an understanding of how experiences during the COVID-19 pandemic (e.g., exposure, risk factors, testing, isolation, seropositivity, hospitalization, loss of family or friends, loss of income), may impact multiple domains of health-related quality of life (physical, emotional and social well-being), and other areas such as COVID-19-specific psychological distress (e.g., fear, anxiety and depressive symptoms), and disruptions to health care, finances, and social interactions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess experiences during the coronavirus disease 2019 (COVID-19) pandemic (e.g., exposure, risk factors, testing, isolation, seropositivity, hospitalization, loss of family or friends); COVID-19-specific psychological distress (e.g., fear, anxiety and depressive symptoms); health, financial and social disruptions; perceived benefits and social support; and health-related quality of life (HRQoL) in a convenience sample of cancer patients and survivors.

II. Evaluate the extent to which COVID-19 experiences are associated with COVID-19-specific psychological distress, health, financial and social disruptions, perceived benefits and social support, and HRQoL.

III. Evaluate the extent to which resiliency factors such as social support and perceived benefits moderate the effects of COVID-19 experiences on COVID-19-specific psychological distress and HRQoL.

OUTLINE:

Patients complete an online questionnaire over 10 minutes regarding the COVID-19 pandemic including testing, risks of exposure, whether people they know have acquired COVID-19, as well as questions on how the pandemic has impacted their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* MD Anderson active patient (visit within past 5 years)
* ICD-10 confirmed cancer diagnosis
* Documentation of being alive per the cancer registry
* Patients who have signed consent for one of the following protocols: PA14-0241 or LAB03-0320
* Has an active email address and/or can be contacted via MyChart
* English or Spanish speaker

Exclusion Criteria:

* Non-active patient (i.e., no visit within past 5 years)
* Language other than English or Spanish
* Patients who have previously consented to the following protocols: 2012-0112, 2009-0976, 2005-0035, or PA15-0336, because they will be contacted through separate IRB protocols to complete this same survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a confirmed cancer diagnosis and cancer survivors
Sampling Method: Non-Probability Sample
Enrollment: 13378 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Experiences during the coronavirus disease 2019 (COVID-19) pandemic | 2 months
  This will be measure with a COVID-19 questionnaire created to collect COVID-19 experience information, Quality of life (QOL), and other psychosocial variables from participating patients. Using this questionnaire may help researchers gain an understanding of how experiences during the COVID-19 pandemic (e.g., exposure, risk factors, testing,isolation,seropositivity, hospitalization, loss of family or friends, loss of income), may impact multiple domains of health-related quality of life (physical, emotional and social well-being), and other areas such as COVID-19-specific psychological distress (e.g., fear, anxiety and depressive symptoms), and disruptions to health care, finances, and social interactions.
COVID-19-specific psychological distress | Up to 2 months
  This will be measure with a COVID-19 questionnaire created to collect COVID-19 experience information, Quality of life (QOL), and other psychosocial variables from participating patients. Using this questionnaire may help researchers gain an understanding of how experiences during the COVID-19 pandemic (e.g., exposure, risk factors, testing,isolation,seropositivity, hospitalization, loss of family or friends, loss of income), may impact multiple domains of health-related quality of life (physical, emotional and social well-being), and other areas such as COVID-19-specific psychological distress (e.g., fear, anxiety and depressive symptoms), and disruptions to health care, finances, and social interactions.
COVID-19-specific health | Up to 2 months
  This will be measure with a COVID-19 questionnaire created to collect COVID-19 experience information, Quality of life (QOL), and other psychosocial variables from participating patients. Using this questionnaire may help researchers gain an understanding of how experiences during the COVID-19 pandemic (e.g., exposure, risk factors, testing,isolation,seropositivity, hospitalization, loss of family or friends, loss of income), may impact multiple domains of health-related quality of life (physical, emotional and social well-being), and other areas such as COVID-19-specific psychological distress (e.g., fear, anxiety and depressive symptoms), and disruptions to health care, finances, and social interactions.
COVID-19-specific financial and social disruptions | Up to 2 months
  This will be measure with a COVID-19 questionnaire created to collect COVID-19 experience information, Quality of life (QOL), and other psychosocial variables from participating patients. Using this questionnaire may help researchers gain an understanding of how experiences during the COVID-19 pandemic (e.g., exposure, risk factors, testing,isolation,seropositivity, hospitalization, loss of family or friends, loss of income), may impact multiple domains of health-related quality of life (physical, emotional and social well-being), and other areas such as COVID-19-specific psychological distress (e.g., fear, anxiety and depressive symptoms), and disruptions to health care, finances, and social interactions.
COVID-19-specific perceived benefits and social support | Up to 2 months
  This will be measure with a COVID-19 questionnaire created to collect COVID-19 experience information, Quality of life (QOL), and other psychosocial variables from participating patients. Using this questionnaire may help researchers gain an understanding of how experiences during the COVID-19 pandemic (e.g., exposure, risk factors, testing,isolation,seropositivity, hospitalization, loss of family or friends, loss of income), may impact multiple domains of health-related quality of life (physical, emotional and social well-being), and other areas such as COVID-19-specific psychological distress (e.g., fear, anxiety and depressive symptoms), and disruptions to health care, finances, and social interactions.
COVID-19-specific health related quality of life (HRQoL) | Up to 2 months
  This will be measure with a COVID-19 questionnaire created to collect COVID-19 experience information, Quality of life (QOL), and other psychosocial variables from participating patients. Using this questionnaire may help researchers gain an understanding of how experiences during the COVID-19 pandemic (e.g., exposure, risk factors, testing,isolation,seropositivity, hospitalization, loss of family or friends, loss of income), may impact multiple domains of health-related quality of life (physical, emotional and social well-being), and other areas such as COVID-19-specific psychological distress (e.g., fear, anxiety and depressive symptoms), and disruptions to health care, finances, and social interactions.
Effects of COVID-19 experiences on COVID-19-specific psychological distress and HRQoL | Up to 2 months
  Will evaluate the extent to which resiliency factors such as social support and perceived benefits moderate the effects of COVID-19 experiences on COVID-19-specific psychological distress and HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org